CLINICAL TRIAL: NCT04216732
Title: Utilization of the Natural History of Medullary Thyroid Carcinoma to Inform Advanced Disease Management
Brief Title: Natural History of Medullary Thyroid Cancer to Inform Advanced Disease Management
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-0769; NCI-2019-07526 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0769 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-14; First posted 2020-01-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Advanced Thyroid Gland Medullary Carcinoma; Stage III Thyroid Gland Medullary Carcinoma AJCC v8; Stage IV Thyroid Gland Medullary Carcinoma AJCC v8; Stage IVA Thyroid Gland Medullary Carcinoma AJCC v8; Stage IVB Thyroid Gland Medullary Carcinoma AJCC v8; Stage IVC Thyroid Gland Medullary Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, blood pressure): AIM I & II: Patients complete questionnaires over 10-40 minutes 2-4 times per year about health and how finances and quality of life effect experience with disease.
  AIM III: Patients complete a questionnaire over 2 minutes and undergo blood pressure measurements every day for up to 12 weeks.
  Interventions: Other: Blood Pressure Measurement; Other: Questionnaire Administration

INTERVENTIONS:
Other: Blood Pressure Measurement — Undergo blood pressure measurement
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study utilizes a multi-institutional registry to describe the natural history of medullary thyroid cancer that has spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) in understanding disease management. The goal of this study is to learn about how medullary thyroid cancer develops and progresses.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the natural history of medullary thyroid cancer (MTC) using a comprehensive battery of demographic, clinical, pathologic, and genotypic variables collected in our existing multi-institutional patient registry.

Ia. To describe the demographic, clinical, pathologic, and genotypic variables associated with each phase of disease.

Ib. To identify those variables which are predictors of progression to the most advanced phases of disease that require small molecule therapy, including commercially approved and experimental agents.

II. To characterize patients' experience with the different phases of MTC through a systematic evaluation of patient-reported outcomes (PROs).

IIa. To describe clinical, psychosocial, economic, and physical well-being variables and the subsequent impact on quality of life associated with each phase of disease.

IIb. To evaluate longitudinal changes in clinical, psychosocial, economic, and physical well-being variables between and within all phases of MTC, and the subsequent impact they have on quality of life.

III. To evaluate the association of selected biometric and patient-reported outcomes on adherence, change, and discontinuation of approved targeted therapies and drugs being tested within clinical trial.

OUTLINE:

AIM I & II: Patients complete questionnaires over 10-40 minutes 2-4 times per year about health and how finances and quality of life effect experience with disease.

AIM III: Patients complete a questionnaire over 2 minutes and undergo blood pressure measurements every day for up to 12 weeks.

The questionnaire data gets paired with the collected medical record history that is maintained in the Registry.

ELIGIBILITY:
Inclusion Criteria:

* Aims 1 and 2: A diagnosis of MTC
* Aims 1 and 2: A registrant in the Medullary Thyroid Cancer Registry (MTCR). Patients of all disease phases will be eligible for enrollment
* Aim 3: A diagnosis of advanced phase (red or gray) MTC as determined by clinical team
* Aim 3: A current registrant in the MTCR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with MTC including advanced phase MTC determined by clinical team
Sampling Method: Non-Probability Sample
Enrollment: 2030 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Natural history of medullary thyroid cancer (MTC) | Up to 4 years
  Will describe the natural history of MTC using comprehensive battery of demographic, clinical, pathologic, and genotypic variables collected in existing multi-institutional patient registry.
Patients' experience with the different phases of MTC | Up to 4 years
  Will characterize patients' experience with the different phases of MTC through a systematic evaluation of patient-reported outcomes (PROs).
Association of selected biometric and patient-reported outcomes | Up to 4 years
  Will evaluate the association of selected biometric and patient-reported outcomes on adherence, change, and discontinuation of approved targeted therapies and drugs being tested within clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G Grubbs, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: http://www.mdanderson.org — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-09-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT04216732/ICF_001.pdf